CLINICAL TRIAL: NCT03247413
Title: Post-lesion Administration of Dexamethasone to Prevent the Development of Neuritis After Radiofrequency Ablation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has been halted prematurely
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00113297
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Neuritis; Radiofrequency Ablation
MeSH Terms: conditions — Neuritis | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Each patient serves as his or her own control. Investigators are recruiting patients who are undergoing bilateral procedures. Each patient will receive dexamethasone at each lesion site post-ablation on one side, and placebo (saline) on the other.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, care providers, and principle investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Lesions where dexamethasone 4 milligram is administered post-radiofrequency ablation
  Interventions: Drug: Dexamethasone 4 mg/ml
- Placebo (Placebo Comparator): Lesions where 1 milliliter of normal saline is administered post-radiofrequency ablation
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone 4 mg/ml — dexamethasone 4 milligram given post-ablation at each lesion site
  Arms: Dexamethasone
Drug: Normal saline — Placebo, normal saline administered post-ablation at each lesion site
  Arms: Placebo

SUMMARY:
Chronic neck and back pain has become one of the leading causes of disability and loss of productivity. For many patients with facet or sacroiliac joint mediated pain who have responded to diagnostic nerve blocks, radiofrequency ablation of the nerves innervating the joints can provide long term relief. Radiofrequency ablation (RFA) is a relatively safe procedure with minimal risk of adverse events. However, with any procedure involving damage to the peripheral nervous system, there is risk of post-procedure neuropathic pain. The investigators will test the hypothesis that dexamethasone injection delivered at the time of lesion effectively prevents the development of post-ablation neuritis through a placebo-controlled, double-blind, randomized trial in patients undergoing cervical, thoracic, lumbar, and sacroiliac joint radiofrequency denervations

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of either cervical, thoracic, or lumbar facet or sacroiliac joint pain who have responded to medial branch blocks and are already scheduled for bilateral radiofrequency ablations
* age greater than 18 years old
* English speaking

Exclusion Criteria:

* patient not previously scheduled for radiofrequency ablation of the cervical, thoracic, or lumbar facets, or sacroiliac joints
* on anticoagulation
* have a pacemaker
* age less than 18 years old
* non-English speaking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Chhatre, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Result] Shustorovich A, AlFarra T, Arel AT, Singh JR, Roemmich RT, Chhatre A. Dexamethasone Effectively Reduces the Incidence of Post-neurotomy Neuropathic Pain: A Randomized Controlled Pilot Study. Pain Physician. 2021 Dec;24(8):517-524. PMID 34793638

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Groups:
- All Study Participants: Each patient received both the dexamethasone and placebo on alternating sides of the affected spinal level.
  One Lesion where dexamethasone 4 milligram is administered post-radiofrequency ablation Dexamethasone 4 mg/ml: dexamethasone 4 milligram given post-ablation at each lesion site On the opposing side, 1 milligram of normal saline was given.
Period: Overall Study
Arm/Group | All Study Participants
Started | 63; 126 Lesions
Received Dexamethasone (4 mg/ml) Intervention | 63; 126 Lesions
Received Placebo (1 mg Saline) Intervention | 63; 126 Lesions
Completed | 35; 70 Lesions
Not Completed | 28; 56 Lesions
Not completed — Lost to Follow-up | 28

BASELINE CHARACTERISTICS:
Groups:
- Dexamethasone/Placebo: Each patient received bilateral lesions on either side of the spinal level and served as their own control arm.
  Lesions where dexamethasone 4 milligram is administered post-radiofrequency ablation
  Dexamethasone 4 mg/ml: dexamethasone 4 milligram given post-ablation at each lesion site
  Lesions where 1 milliliter of normal saline is administered post-radiofrequency ablation
  Normal saline: Placebo, normal saline administered post-ablation at each lesion site
Arm/Group | Dexamethasone/Placebo
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35
Post-neurotomy pain incidence [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With Post-Ablation Neuritis
Description: Each patient had 2 lesions. One Lesion was treated with dexamethasone. The other lesion was treated with placebo. We then looked at the number of lesions that developed post-ablation neuritis.
Time Frame: 4 weeks
Measure: Number; unit: lesions
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 35 | 35
lesions | 3 | 20

ADVERSE EVENTS:
Time Frame: 1 year
Description: 35 participants of the original 63 that were enrolled participated in the study and were at risk of adverse events.
Groups:
- Dexamethasone/Placebo: Each patient received both the dexamethasone and placebo on alternating sides of the spinal level.
  One Lesions where dexamethasone 4 milligram is administered post-radiofrequency ablation Dexamethasone 4 mg/ml: dexamethasone 4 milligram given post-ablation at each lesion site On the opposing side, 1 milligram of normal saline was given
Arm/Group | Dexamethasone/Placebo
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT03247413/Prot_SAP_000.pdf